CLINICAL TRIAL: NCT02637089
Title: Longitudinal Comparison of the Nature and Evolution of Mild Cognitive Impairment in Individuals With and Without Parkinson's Disease Characterized by Neuroimaging, Clinical Assessments and Genotyping
Brief Title: Longitudinal Study of Mild Cognitive Impairment in Parkinson's Disease
Acronym: PD-MCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Natural Sciences and Engineering Research Council, Canada (Other); Montreal Neurological Institute and Hospital (Other); McGill University (Other)
Responsible Party: Principal Investigator, Oury Monchi, Professor, University of Calgary
Other Study IDs: REB14-2463
Record Dates: First submitted 2015-09-09; First posted 2015-12-22 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Parkinson's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 60 ml of blood will be collected from all participants to analyze biomarkers and DNA for genes of interest
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- PD-non-MCI: Patients with Parkinson's disease, no mild cognitive impairment
- PD-MCI: Patients with Parkinson's disease with mild cognitive impairment
- MCI (non-PD-MCI): Patients with mild cognitive impairment, no Parkinson's disease
- HC (non-PD-non-MCI): Healthy Controls (age-matched to patients)

SUMMARY:
Parkinson's disease (PD) is known for its motor symptoms and affects more than 100,000 Canadians. However, PD patients also show cognitive deficits and neuropsychiatric problems that significantly impair their quality of life. The occurrence of dementia in PD is much higher than in the general population. The proposed study will allow the principal investigator, his team and his collaborators to investigate the origins and evolution of the cognitive and neuropsychiatric symptoms. Participants with PD with and without mild cognitive impairment (MCI) and participants with and without MCI over the age of 60 years will be assessed during eight study visits over three years. Through brain imaging, clinical testing, as well as genotyping the cognitive patterns in the four different groups will be observed and compared. The results will be used to identify biomarkers that can predict the occurrence of dementia early in the disease. Ultimately, the results of the proposed research will contribute to interventions and treatment strategies tailored to different cognitive profiles in PD before the occurrence of dementia.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most frequent chronic neurodegenerative disorder, affecting up to 2% among persons older than 65 years of age and nearly 10% of people over 80. The cardinal symptoms of PD include tremor, rigidity and bradykinesia originating from the loss of dopaminergic neurons in the striatum. It has recently been shown that the non-motor symptoms in PD such as cognitive and behavioural impairment are highly prevalent and have a severe and direct negative effect on health-related and perceived quality of life. It is now well established that 25 to 40% of persons with PD will develop cognitive deficits early in the disease. Moreover, the risk of developing dementia is almost six times higher in PD patients than in age-matched controls. The nature and evolution of cognitive deficits in PD remain poorly understood, so is their relationship with neuropsychiatric features often observed in the disease including depression, anxiety and apathy. Furthermore, the medication treatment of cognitive deficits in PD yields very modest results. PD neuropathology is associated with alpha-synuclein-containing Lewy-Bodies whereas that of Alzheimer's disease (AD) is usually associated with Aß-amyloid plaques and tau-containing neurofibrillary lesions. However, recent post-mortem studies suggest that between 30 and 45% of PD patients with dementia also meet neuropathologic diagnostic criteria for AD. With such a high proportion of demented PD patients with concurrent AD, it would be valuable, from a therapeutic standpoint, to identify those with AD earlier. In the context of the present proposal the investigators will be able to follow different groups of PD patients longitudinally and compare them to non-PD patients with mild cognitive impairment who are at risk of developing a medio-temporal lobe dementia such as Alzheimer's disease.

The three major aims for this longitudinal study are:

1. Identify anatomical and functional neuroimaging, neuropsychological and neuropsychiatric profiles that can serve as markers for the early prediction of dementia in PD.
2. Uncover the cognitive and neural characteristics that are specific to PD-MCI subjects vs. characteristics shared by all MCI subjects whether due to PD or other aetiology such as Alzheimer's disease.
3. Identify the effect of specific genotypes that can influence the cognitive profile and evolution in PD.

The investigators will recruit 100 PD and 100 non-PD individuals. None of them will have dementia. Participants will be selected in order to obtain about 65% MCI and 35% cognitively intact individuals in each cohort (PD, non-PD). At study start they will be asked to consent to a blood draw for genotyping purposes. At each time point, they will receive a neuropsychological evaluation to determine whether and which domain(s) of cognition is (are) affected and whether the participant meets the criteria for dementia. Neuropsychiatric symptoms which are often present before the onset of cognitive symptoms will be assessed at each time point using the Mild Behavioural Impairment-Checklist (MBI-C). At Time points 1 and 2 they will also undergo two MRI sessions containing anatomical acquisitions as well as BOLD functional series while performing an executive (set-shifting) task that the investigators have shown to rely on fronto-striatal regions and an (associative) memory task that solicits the medial temporal lobe. At Time point 3 they will undergo just one MRI session not containing any task. This will allow the investigators to identify markers that can distinguish subgroups with respect to their possible evolution towards dementia. This multi-faceted, longitudinal project promises to enhance the understanding of the nature and evolution of cognitive dysfunction in PD relative to general aging. To the investigators' knowledge, this is the first time that PD and non-PD patients stratified according to cognitive profile will be studied longitudinally using neuropsychological evaluation, anatomical and functional neuroimaging measures as well as genotyping. This information has the potential to yield markers that can be used in clinics to determine the diagnosis and prognosis of cognitive dysfunction in PD, allowing for an early prediction of dementia in the disease. This will ultimately yield intervention and treatment strategies tailored to different patient subtypes, aimed at improving cognitive deficits and decelerating the decline.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Non-demented PD patients at stages II or III of Hoehn and Yahr at Time point 1 with or without MCI
* MCI patients
* Willing and able to provide written informed consent
* Willing to provide blood sample, willing to participate in all clinical assessments, willing to have brain MRIs

Controls:

* Community volunteers, with no history of PD or cognitive or memory complaints
* Willing and able to provide written informed consent
* Willing to provide blood sample, willing to participate in all clinical assessments, willing to have brain MRIs
* Screen negative for MCI

Exclusion Criteria:

•All participants who meet the diagnosis of dementia at Time point 1 as indicated by Mini-Mental State Evaluation (MMSE) of 20 or less and indicated through the clinical testing.

(The neuropsychological evaluation will always take place before the imaging sessions, in case participants must be excluded based on their cognitive profile.)

* All participants taking benzodiazepines will be excluded as these can severely impair performance of cognitive tasks.
* Participants with metallic objects in their bodies will not be eligible for the study because the strong magnetic field in the scanner could cause these objects to change position and may cause injury.
* The following criteria will also be used as grounds for exclusion, as they have severe impact on cognitive function:

  * Alcohol-dependency
  * Presence or history of severe psychiatric disorder, neurological disorder or stroke
  * General anaesthesia in the past six months
  * History of cerebrovascular disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease with and without mild cognitive impairment, patients without Parkinson's disease with and without (healthy controls) mild cognitive impairment, 60 years of age or older
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-03-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Identify which structures in the brain exhibit the highest structural changes and / or BOLD changes correlated to the Z-scores of the neuropsychological assessments | Baseline, 18 months, 36 months
  Structural changes and changes in BOLD fMRI sequence will be measured at each of the three time points. These measurements will be correlated to the Z-scores of the neuropsychological assessments at each time point.

SECONDARY OUTCOMES:
Change from baseline in Z-scores of different neuropsychological assessments | Baseline, 18 months, 36 months
  1. Change in Z-scores overall
  2. Change in Z-scores per domain:
  Executive, Attention, Visio-spatial and Visio-perceptual, Language, Verbal and Episodic Memory and Global Cognition
Change in Cognitive Ability measured as BOLD fMRI sequence | Baseline, 18 months, 36 months
  Establish an episodic imaging memory task to be performed in the scanner to measure the level of medial temporal lobe activation via BOLD fMRI sequence (blood-oxygen-level-dependent contrast imaging)
Change in Executive Functioning measured as BOLD fMRI sequence | Baseline, 18 months, 36 months
  Establish an executive task to be performed in the scanner to measure the level of activation in the basal ganglia and the prefrontal cortex via BOLD fMRI sequence (blood-oxygen-level-dependent contrast imaging)
Measure changes in the volume of subcortical structures in the brain | Baseline, 18 months, 36 months
  Volume of subcortical structures (mm3)
Measure changes in cortical thickness in the brain | Baseline, 18 months, 36 months
  Cortical thickness (mm)
Measure structural changes in the brain | Baseline, 18 months, 36 months
  Rate of change in cortical thickness (mm/year)
Analyze DNA for following genes: COMT, DAT1, MAPT, ApoE, GBA, CHNRA4 | Baseline
  Genotyping
Measure level of biomarkers: Aß-amyloid in blood through fluorescence spectroscopy | Baseline
  Increase or decrease in fluorescence can be determined visually by looking at spectral fluorescence images. Increased fluorescence can be quantified in % compared to blood from a participant who has no disease associated with abnormal protein aggregation.
Measure psychiatric changes with the Mild Behavioural Impairment-Checklist (MBI-C) | Baseline, 18 months, 36 months
  Changes in scores per domain

CONTACTS AND LOCATIONS:
Overall Officials: Oury Monchi, PhD, Principal Investigator — University of Calgary, Cumming School of Medicine, Department of Clinical Neurosciences
Locations (1):
- University of Calgary, Department of Clinical Neurosciences, Calgary, Alberta, Canada